CLINICAL TRIAL: NCT03253978
Title: A Randomised Feasibility Study Evaluating Stereotactic Prostate Radiotherapy In High-Risk Localised Prostate Cancer With or Without Elective Nodal Irradiation
Brief Title: SPORT High-Risk Trial Evaluating SABR in Prostate Cancer
Acronym: SPORT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14190SJ-SS
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: A randomised feasibility study
Masking Description: Not applicable - no masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SABR to prostate / seminal vesicles with pelvic ENI (Experimental): 36.25Gy / 5 fractions to prostate and seminal vesicles with additional SABR (25Gy /5 fractions) delivered to the pelvic nodes.
  Interventions: Radiation: Stereotatic Radiotherapy
- SABR to prostate and seminal vesicles only (Active Comparator): 36.25Gy / 5 fractions to prostate and seminal vesicles.
  Interventions: Radiation: Stereotatic Radiotherapy

INTERVENTIONS:
Radiation: Stereotatic Radiotherapy — SABR to prostate / seminal nodes

SUMMARY:
The study will examine stereotactic ablative body radiotherapy (SABR), a new technique to deliver radiotherapy to men with prostate cancer. In addition to this, it will look at the effect of SABR on levels of markers of radiation exposure and bowel damage, along with other potential markers of outcome and side effects. Quality of life and any side effects that develop during and after treatment will also be assessed.

DETAILED DESCRIPTION:
The study will examine stereotactic ablative body radiotherapy (SABR), a new technique to deliver radiotherapy to men with prostate cancer. In addition to this, it will look at the effect of SABR on levels of markers of radiation exposure and bowel damage, along with other potential markers of outcome and side effects. Quality of life and any side effects that develop during and after treatment will also be assessed.

Participants will be treated with five treatments (instead of the standard 37). This is more convenient for them and also allows the treatment of many more people in the same time frame, which should improve the timely delivery of radiotherapy for all patients.

Thirty men with high-risk prostate cancer will be enrolled into the study. They will all be treated with hormone therapy and radiotherapy to the prostate and seminal vesicles. In addition, half of the men will receive an additional dose of radiation to their pelvis. Gold markers will be placed in the prostate before radiotherapy to allow precise targeting of the prostate during treatment. CT scans are taken before and after each treatment to ensure the accuracy of its delivery.

Blood urine and prostate tissue samples will be taken before, during and after radiotherapy. Side effects and quality of life will also by assessed during this time.

Ultimately, this may allow us to predict which men are at increased risk of side effects from radiotherapy and allow closer monitoring, earlier intervention and perhaps alternative treatments in some cases. This should improve the control of prostate cancer and reduce the risk of serious treatment-related side effects

ELIGIBILITY:
Inclusion Criteria:

Patients with histologically confirmed prostate adenocarcinoma who elect for radical radiotherapy, with at least one of the following features:

* clinical stage T3a N0 M0
* Gleason score 7 (4+3) or above
* PSA > 20

No evidence of nodal or distant metastatic disease

WHO performance status 0-2

Life expectancy of at least 5 years

Men greater than or equal to 18 years

Ability to understand and willingness to sign a written informed consent document (completed prior to registration and subsequent randomization), along with willingness to co-operate with follow-up

Planned to receive 12-36 months of ADT as part of standard treatment

Exclusion Criteria:

T stage greater than or equal to T3b / T4

Prostate volume > 90cc

Current evidence of:

* inflammatory bowel disease or other chronic bowel disorder
* Autoimmune disease
* Active uncontrolled bacterial, viral or fungal infection
* Serious uncontrolled concomitant disease
* Known coagulopathy or bleeding diasthesis
* Anticoagulation medication (if unsafe to insert for seed insertion)
* Bilateral hip prosthesis or fixation which would interfere with standard radiation beam configuration
* Concurrent experimental or cytotoxic drugs
* Allergy to gold
* Severe lower urinary tract symptoms - International Prostate Symptom Score (IPSS) > 19
* Any other contra-indication to hormonal therapy or radical radiotherapy.

History of:

* Previous major abdominal surgery or history of bowel adhesions
* Prior pelvic radiotherapy
* Active malignancy within the preceding five years (other than basal cell carcinoma)

Evidence of:

- Castrate-resistance (rising PSA with castrate levels of testosterone on LHRHa and anti-androgen)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men with newly diagnosed high-risk localized prostate cancer
Enrollment: 40 (Actual)
Dates: Start 2016-01-18 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Adequate recruitment rate | 24 months
  adequate recruitment rate (30 patients in 24 months)
Acute toxicity of SABR | 90 days of completion of SABR
  Acute toxicity of SABR (as assessed by CTCAE v4.03 scores until 90 days of completion of SABR)
Acute quality of life during and after SABR | 90 days after completion of SABR
  Acute quality of life during and after SABR (as assessed by EPIC and IPSS scores until 90 days after completion of SABR)
Number of SABR plans delivered as planned and on schedule | 29 days (treatment period)
  Number of SABR plans delivered as planned and on schedule
Quantification of acute toxicity in each treatment group | until 90 days post completion of radiotherapy
  Quantification of acute toxicity in each treatment group to enable calculation of the sample size for the Phase II RCT (using CTCAE v4.03 scores measured until 90days post completion of radiotherapy)

SECONDARY OUTCOMES:
Late toxicity of SABR | from 90 days and up to ten years post completion of SABR
  Late toxicity of SABR (as assessed by GI and GU RTOG late toxicity scores from 90 days to ten years post completion of SABR)
Late patient-reported quality of life | up to ten years post completion of SABR
  Late patient-reported quality of life (as assessed by EPIC and IPSS scores from 90 days to ten years post completion of SABR)
Rate of PSA failure | up to ten years post completion of SABR
  Rate of PSA failure as assessed by Phoenix criteria
Prostate cancer-specific survival | up to ten years post completion of SABR
  Prostate cancer-specific survival
Overall survival | up to ten years post completion of SABR
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Suneil Jain, Dr, Principal Investigator — Chief Investigator
Locations (1):
- Belfast Health and Social Care Trust, Belfast, Co. Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We would welcome collaboration with other researchers as long as full ethical approval was granted